

7.1.2019, Version 2.

Clinical Trial unique protocol ID 2017/12883-2

## Invitation to participate in the research project

# "Nutrition and Medication" part II, (Nedre Eiker)

This is an invitation were we ask if you may be willing to be a participant in a research project concerning nutritional status and medication use among elderly persons receiving home nurse services.

Many older adults are not able to get sufficient food intake and are at risk for malnutrition. Adverse medication effects, as reduced appetite, nausea or dry mouth can contribute to malnutrition. The aim of the project is to investigate if an individual tailored nutritional plan and medication review can improve nutritional status, quality of life, functioning in daily living activities, or reduce admissions to hospital or nursing homes. The study is a part of a Ph.D.-project, and the project will be done in collaboration with the Health and Care Services in your home municipality.

### What does participation in the project imply for you?

If you accept to participate, a qualified nurse or another health care worker from the Home Nurse Service will visit you. You will be asked questions about your life situation, nutritional habits, your need for help in daily living activities, and about your own assessment of your health related quality of life. You will be weighed, and a photo of your medication card will be taken. We will ask for your permission to ask your General Practitioner about how many times you eventually have been to a hospital during the last six months and the project period. We will also ask for permission to get information from the Health and Care Services in the municipality about eventually admissions to short time ward in a nursing home during the same period. As part of the project, you will be visited twice in your own home in the beginning of the project period, and after six months.

## Possible benefits and risks by participation

Participating in this project does not imply any risks for you, but you will need to spend approximately 15-20 minutes with us for each of the two visits. If something will be disclosed which probably should be assessed by your doctor, the Home Nursing Service will with your acceptance contact your General Practitioner.

#### Voluntary participation and the possibility to withdraw consent

Participation in the project is voluntary. If you want to participate, you will need to sign the declaration of consent (last page in this letter). At any given time and without need for



# **UiO** "Nutrition and Medication" Part- II, (Nedre Eiker) 7.1.2019, version 2

giving reasons, you are free to withdraw your consent. This will not have any consequences for future provision of health care for you. If you decide to withdraw participation in the project, you are also free to demand that your data file in this project can be deleted, unless if your anonymized data have already been analysed or used in scientific publications.

If you at a later point, wish to withdraw your consent or have any questions regarding the project, you can contact Ph.D.- candidate and nursing home physician Mari Fiske, University of Oslo, mari.fiske@medisin.uio.no, telephone 926 67 311.

## What will happen to your personal data concerning health?

Any personal data concerning health that has been recorded about you, will only be used as described in the purpose for the project. You have the right to access information that has been recorded for you and also the right to see that any error(s) in the recorded data is/ are corrected. You also have the right to know which security measures that have been/will be taken when personal data concerning health is processed.

All information will be processed and used without names or personal identification numbers, or any other information that may directly identify the participants. Linkage between you and your health data will only be possible via a separate identifier list. Only the researchers, professors Jørund Straand, Anne Moen and Ph. D. - candidate and nursing home physician Mari Fiske will have access to the list.

#### **Finance**

The project is funded by The Norwegian Research Fund for General Practice and the County Governor in Buskerud, Norway.

#### **Approval**

The Regional Committee for Medical and Health Research Ethics has reviewed and approved the Research Project. Reference number 2018/1045.

In accordance with the General Data Protection Regulation, the University of Oslo and the project manager, Professor Jørund Straand, is independently responsible for ensuring that the processing of your personal health data has a legal foundation. This project has a legal foundation in accordance with the EU General Data Protection Regulation, article 6 no. 1a, article 9 no. 2a, and with your consent. You have the right to eventually submit a complaint on the processing of personal health data to the Norwegian Data Inspectorate.

#### **Contact information**

If you have any questions regarding the research project, you can get in touch with Mari Fiske, University of Oslo, Email: <a href="mari.fiske@medisin.uio.no">mari.fiske@medisin.uio.no</a>, telephone: 926 67 311 Jørund Straand, University of Oslo, Email: <a href="mailto:jorund.staand@medisin.uio.no">jorund.staand@medisin.uio.no</a>, telephone: 928

# UiO \* "Nutrition and Medication" Part- II, (Nedre Eiker) 7.1.2019, version 2

| 52 | 523; | or |
|----|------|----------|
| J- | J-J, | <b>-</b> |

Anne Moen, University of Oslo, Email: <a href="mailto:anne.moen@medisin.uio.no">anne.moen@medisin.uio.no</a>

I consent to participating in the research project and that my personal data concerning health can be used as described above

| City/Town and date | Participant's Signature |
|--------------------------------------------|------------------------------|
| | Participant's Name (in BLOCK |
| | LETTERS) |
| I confirm that I have given information al | oout the research project |
| City/Town and date | Signature |
| | Role in the research project |